CLINICAL TRIAL: NCT00524732
Title: Assessment of the Reactogenicity of ADACEL® (TdcP Vaccine) in Children and Adolescents 7 to 19 Years of Age
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: TD511
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Pertussis; Diphtheria
Keywords: Pertussis; Tetanus; Diphtheria
MeSH Terms: conditions — Whooping Cough; Diphtheria; Tetanus | interventions — Tetanus Toxoid; adacel

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- 1: 18 to 30 months since last prior dose of TD/Td vaccine.
  Interventions: Biological: Tetanus and diphtheria toxoids and acellular pertussis
- 2: 30 to 42 months since last prior dose of TD/Td vaccine.
  Interventions: Biological: Tetanus and diphtheria toxoids and acellular pertussis
- 3: 42 to 54 months since last prior dose of TD/Td vaccine.
  Interventions: Biological: Tetanus and diphtheria toxoids and acellular pertussis
- 4: 54 to 66 months since last prior dose of TD/Td vaccine.
  Interventions: Biological: Tetanus and diphtheria toxoids and acellular pertussis
- 5: 66 to 78 months since last prior dose of TD/Td vaccine.
  Interventions: Biological: Tetanus and diphtheria toxoids and acellular pertussis
- 6: 78 to 90 months since last prior dose of TD/Td vaccine.
  Interventions: Biological: Tetanus and diphtheria toxoids and acellular pertussis
- 7: 90 to 102 months since last prior dose of TD/Td vaccine.
  Interventions: Biological: Tetanus and diphtheria toxoids and acellular pertussis
- 8: 102 to 114 months since last prior dose of TD/Td vaccine.
  Interventions: Biological: Tetanus and diphtheria toxoids and acellular pertussis
- 9: Control - over 114 months since last prior dose of TD/Td vaccine.
  Interventions: Biological: Tetanus and diphtheria toxoids and acellular pertussis

INTERVENTIONS:
Biological: Tetanus and diphtheria toxoids and acellular pertussis — 0.5 mL, Intramuscular
  Other Names: ADACEL®

SUMMARY:
To compare the reactogenicity of ADACEL® vaccine given at intervals of 2 to 9 years with the reactogenicity of ADACEL® vaccine given at an interval of 10 or more years following the last previous administration of vaccine containing Diphtheria and Tetanus Toxoids (referred to as TD/Td).

ELIGIBILITY:
Inclusion Criteria:

* Age > 7 years and < 20 years.
* Signed and dated IRB-approved informed consent form obtained from the participant, parent or legal guardian prior to the first study intervention.
* Judged to be in good health on the basis of reported medical history.
* Available for planned length of the study.
* Participant or parent or legal guardian (as applicable) can read and write English and can understand the informed consent documents and the study instructions.

A participant eleven years of age or older who meets an exclusion criterion may not be enrolled in the study but nonetheless may participate in the vaccination program, at the discretion of the Prince Edward Island public health authorities).

A participant younger than eleven years of age who meets an exclusion criterion may not be enrolled in the study and may not participate in the vaccination program.

Exclusion Criteria:

* Known or suspected allergy to ADACEL®, any of the vaccine's components, or prior allergic reaction to Diphtheria or Tetanus Toxoids or Acellular Pertussis Vaccine.
* Planned receipt of any other vaccine within the 14 days following administration of ADACEL® vaccine in this study.
* Any other medical condition that in the opinion of the investigator would cause an unexpected hazard or interfere with the study objective.
* Receipt of TD/Td within the preceding 12 months.
* Known or suspected to be pregnant.

A participant eleven years of age or older who meets an exclusion criterion may not be enrolled in the study but nonetheless may participate in the vaccination program, at the discretion of the Prince Edward Island public health authorities).

A participant younger than eleven years of age who meets an exclusion criterion may not be enrolled in the study and may not participate in the vaccination program.

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and Adolescents 7 to 19 Years of Age, who have previously recieved Tetanus and Diphtheria Toxoids Vaccine
Sampling Method: Non-Probability Sample
Enrollment: 7156 (Actual)
Dates: Start 2004-09; Primary Completion 2004-12 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To provide safety information on ADACEL® vaccine given at different time intervals. | Up to 114 months post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Canada (2):
  - Halifax, Nova Scotia
  - Charlottetown

REFERENCES:
- [Result] Halperin SA, Sweet L, Baxendale D, Neatby A, Rykers P, Smith B, Zelman M, Maus D, Lavigne P, Decker MD. How soon after a prior tetanus-diphtheria vaccination can one give adult formulation tetanus-diphtheria-acellular pertussis vaccine? Pediatr Infect Dis J. 2006 Mar;25(3):195-200. doi: 10.1097/01.inf.0000202082.56403.c4. PMID 16511379
- See also: Related Info — http://www.sanofipasteur.com